CLINICAL TRIAL: NCT05047783
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate the Anti-viral Efficacy of Masitinib in Patients With Symptomatic Mild to Moderate COVID-19
Brief Title: Masitinib in Patients With Symptomatic Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB21002; 2021-002620-20 (EudraCT Number)
Record Dates: First submitted 2021-09-16; First posted 2021-09-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Covid19; SARS-CoV2 Infection; Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — masitinib

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Masitinib 3.0 mg/kg/day (Experimental): Masitinib 3.0 mg/kg/day for 10 days versus corresponding placebo (all patients will receive Best Supportive Care)
  Interventions: Drug: Masitinib Mesylate
- Masitinib 4.5 mg/kg/day (Experimental): Masitinib 3.0 mg/kg/day for 2 days then 4.5 mg/kg/day for 8 days versus corresponding placebo (all patients will receive Best Supportive Care)
  Interventions: Drug: Masitinib Mesylate
- Masitinib 6.0 mg/kg/day (Experimental): Masitinib 3.0 mg/kg/day for 2 days then 4.5 mg/kg/day for 2 days then 6.0 mg/kg/day for 6 days versus corresponding placebo (all patients will receive Best Supportive Care)
  Interventions: Drug: Masitinib Mesylate
- Placebo (Placebo Comparator): Placebo arms associated with the three Experimental arms (all patients will receive Best Supportive Care) which will be pooled for analysis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib Mesylate — 3CL-protease inhibitor
  Other Names: Masitinib; AB1010
  Arms: Masitinib 3.0 mg/kg/day; Masitinib 4.5 mg/kg/day; Masitinib 6.0 mg/kg/day
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the anti-viral efficacy of 3 different dosages of masitinib in patients with symptomatic mild to moderate COVID-19.

DETAILED DESCRIPTION:
The primary objective is to evaluate the virologic efficacy of masitinib plus Best Supportive Care (BSC), with respect to placebo plus BSC in reducing viral shedding of SARS-CoV-2 in patients with symptomatic mild to moderate COVID-19.

Patients will be randomized into one of the following treatment groups (all patients will receive BSC):

1. Masitinib 3.0 mg/kg/day for 10 days versus corresponding placebo
2. Masitinib 3.0 mg/kg/day for 2 days then 4.5 mg/kg/day for 8 days versus corresponding placebo
3. Masitinib 3.0 mg/kg/day for 2 days then 4.5 mg/kg/day for 2 days then 6.0 mg/kg/day for 6 days versus corresponding placebo Treatments will be administered for 10 days and patients will be followed for 1 month. The treatment groups will be compared to pooled placebo after unblinding.

Regarding Best Supportive Care, for patients with a score of 2 and 3 (ambulatory) on the 10-score WHO clinical progression scale, Best Supportive Care is best available therapy in the country at the choice of the investigator excluding any antiviral treatment whether indirect (Ribavirin, Hydroxychloroquine or Chloroquine) or direct (anti-polymerase or antiprotease, including lopinavir/ritonavir fixed dose combination), other investigational treatments for SARS-CoV-2, plasma from a person who recovered from COVID-19, monoclonal antibody therapies and vaccine. For patients with a score of 4 and 5 (hospitalized) on the 10-score WHO clinical progression scale, Best Supportive Care is dexamethasone.

ELIGIBILITY:
Key Inclusion Criteria:

- Male or non-pregnant female with: A. Symptomatic ambulatory male or non-pregnant female adult ≥ 18 years of age at time of enrolment with mild COVID-19 with score 2 or 3 of the 10-score WHO clinical progression scale OR B. Hospitalized male or non-pregnant female adult ≥ 18 years of age at time of enrolment with COVID-19 with score 4 or 5 of the 10-score WHO clinical progression scale.

* Symptoms consistent with COVID-19, as determined by investigator, with onset ≤5 days before randomization
* Positive test for COVID-19 ≤72 hours prior to randomization
* Negative test for the IgG anti-SARS-CoV-2

Key Exclusion Criteria:

* Any use of anti-viral medications up to 7 days before participating in the study
* Receipt of plasma from a person who recovered from COVID-19 (convalescent plasma) any time before participating in the study
* Receipt of last recommended dose of a SARS-CoV-2 vaccine up to 30 days before participating in the study
* Receipt of a monoclonal antibodies up to 30 days before participating in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
SARS-Cov-2 Viral Load at Day 10 | Baseline to Day 10
  Time-weighted average change from baseline in viral shedding

SECONDARY OUTCOMES:
SARS-Cov-2 Viral Load to post-baseline study days | Baseline up to Day 28
  Time-weighted average change from baseline in viral shedding
Time to negative RT-qPCR result | Baseline up to Day 28
  Time to negative RT-qPCR result in all tested samples with no subsequent positive RT-qPCR in any tested samples

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LAURICHESSE, MD, Principal Investigator — CHU Gabriel-Montpied, Clermont-Ferrand
Locations (6):
- Intensive Care Unit, CHU Gabriel-Montpied, Clermont-Ferrand, France
- Russia (3):
  - Gabrichevsky Institute of Epidemiology and Microbiology, Moscow
  - Scientific Research Center Eco-Safety, Saint Petersburg
  - City Clinical Hospital No. 14, Yekaterinburg
- South Africa (2):
  - Netcare Jakaranda Hospital, Pretoria, Gauteng
  - Langeberg Clinical Trials, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No
Masitinib is under clinical investigation and has not yet been approved in any sought-after indication by any health authority worldwide. As such, there is no plan for data-sharing at this point in time.

REFERENCES:
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877